CLINICAL TRIAL: NCT03661034
Title: Multi-Center Study of Tolerability, Safety and Efficacy of Sensory Stimulation at Multiple Dose Levels to Improve Brain Function (Etude Study)
Brief Title: Study of Tolerability, Safety and Efficacy of Sensory Stimulation at Multiple Dose Levels to Improve Brain Function (Etude Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cognito Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-0004
Record Dates: First submitted 2018-08-01; First posted 2018-09-07 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease, Early Onset; Alzheimer Disease; Alzheimer Dementia; Mild Cognitive Impairment; Memory Disorders; Memory Loss; Memory Impairment; Memory Disorders, Age Related; Alzheimer Disease, Late Onset; Cognitive Impairment; Dementia, Mild; Dementia, Alzheimer Type; Cognitive Decline
Keywords: Dementia; Alzheimer's Disease; Memory Loss
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Memory Disorders; Dementia; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Multi-center, four-arm prospective dose-adjusting study (2 cohorts sequentially enrolled, each with 2 randomly assigned dose levels)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Cohort 1, Arm A (Experimental): Dosing 1 hour session per day with GammaSense Stimulation System (non-invasive, non-significant risk)
  Interventions: Device: GammaSense Stimulation System (non-invasive, non-significant risk)
- Cohort 1, Arm B (Experimental): Dosing 1 hour session twice per day with GammaSense Stimulation System (non-invasive, non-significant risk)
  Interventions: Device: GammaSense Stimulation System (non-invasive, non-significant risk)
- Cohort 2, Arm C (Experimental): Dosing 1 hour session every other day or one 2 hour session per day, depending on Interim Analysis outcomes with GammaSense Stimulation System (non-invasive, non-significant risk)
  Interventions: Device: GammaSense Stimulation System (non-invasive, non-significant risk)
- Cohort 2, Arm D (Experimental): Dosing 30 minute session twice per day or 120 minute session twice per day, depending on Interim Analysis outcomes with GammaSense Stimulation System (non-invasive, non-significant risk)
  Interventions: Device: GammaSense Stimulation System (non-invasive, non-significant risk)

INTERVENTIONS:
Device: GammaSense Stimulation System (non-invasive, non-significant risk) — Non-invasive, non-significant risk audio-visual sensory stimulation device
  Other Names: FG-0003

SUMMARY:
The Etude Study is a multi-center, four-arm prospective dose-adjusting study designed to assess the tolerability, safety and efficacy of non-invasive sensory stimulation for patients with cognitive impairment.

DETAILED DESCRIPTION:
Subjects will be enrolled in two Cohorts (N=10 each, enrolled sequentially), and each will assess two different dose levels (randomly assigned). Based on initial outcomes in Cohort 1 at Interim Analysis, the doses for Cohort 2 will be escalated or decreased. Subjects will participate in 1 year (48 weeks) of daily therapy dose using the non-invasive, non-significant risk sensory stimulation medical device.

ELIGIBILITY:
Inclusion Criteria:

* >= 50 Years Old
* MMSE 24 - 30
* Prodromal Alzheimer's Disease (AD), AD or Mild Cognitive Impairment (MCI) due to AD
* Participation of a caregiver / care partner
* Amyloid Positive PET Scan

Exclusion Criteria:

* Profound hearing or visual impairment
* Seizure Disorder
* Use of memantine (Namenda or Namzaric)
* Implantable devices (non-MR compatible)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Amyloid Positron Emission Tomography (PET) Scan | PET Imaging at Baseline, 6 weeks and every 3 months throughout therapy (0, 1.5, 3, 6, 9 and 12 month)
  Movement of amyloid, as measured qualitatively and quantitatively in Amyloid PET Imaging at 0, 1.5, 3, 6, 9 and 12 months following assigned regimen of sensory stimulation treatment sessions
Adverse Events | Over 12 months
  Composite adverse events to be assessed at Interim Analysis (at any point in partial study completion), and final analysis (at 6 and 12 months time points).

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale- Cognitive Subscale (ADAS-Cog) | Baseline, 3, 6, 9 and 12 months
  A scale used to assess cognition; This scale consists of 14 questions assessed resulting in a score from 0 to 90, where a higher score indicates more cognitive disruption.

CONTACTS AND LOCATIONS:
Overall Officials: Evan R Hempel, Study Chair — Cognito Therapeutics
Locations (1):
- Boston Center for Memory, Newton, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No